CLINICAL TRIAL: NCT06210971
Title: Exploratory Study on the Efficacy and Safety of Long-course Neoadjuvant Chemoradiation With Liposomal Irinotecan and Capecitabine Guided by UGT1A1 Status in Patients With Locally Advanced Rectal Cancer
Brief Title: Neoadjuvant Chemoradiation With Nal-IRI and Capecitabine Guided by UGT1A1 Status in Patients With Rectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DEY-CRC-K08
Record Dates: First submitted 2024-01-07; First posted 2024-01-18 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Rectal Cancer
Keywords: UGT1A1; liposomal irinotecan; total neoadjuvant therapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — irinotecan sucrosofate; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liposomal irinotecan-based TNT therapy (Experimental): Concurrent Chemoradiotherapy (Radiation 50.4Gy/28 fractions + Capecitabine 625mg/m^2 bid + Liposomal irinotecan 50mg/m^2) followed by 4-6 cycles of Chemotherapy (Capecitabine 1000mg/m^2 bid d1-7 + Liposomal irinotecan 70mg/m^2 or 50mg/m^2, d1, Q2W) before surgery.
  Interventions: Drug: liposomal irinotecan; Drug: Capecitabine; Radiation: Radiation threapy

INTERVENTIONS:
Drug: liposomal irinotecan — Liposomal irinotecan: 50mg/m^2 or 70mg/m^2
  Other Names: nal-IRI
Drug: Capecitabine — Capecitabine: 625mg/m^2 or 1000mg/m^2 bid.
  Other Names: Xeloda
Radiation: Radiation threapy — 50.4Gy/28 fractions
  Other Names: RT

SUMMARY:
This single-arm trial will explore the efficacy and safety of long-course neoadjuvant chemoradiation with liposomal irinotecan and capecitabine guided by UGT1A1 status in patients with locally advanced rectal cancer.

DETAILED DESCRIPTION:
This is a single-center, single-arm, prospective clinical study. The aim of this study is to explore the short-term and long-term efficacy and safety of total neoadjuvant therapy with irinotecan liposome in patients with locally advanced rectal cancer. Patients' nutritional status, quality of life, changes in symptoms, and adverse events will also be regularly assessed and registered during the implementation phase of the study, and patients will be treated promptly if symptoms are assessed as positive.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18~75 years old.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0~1.
* Histopathologically confirmed rectal adenocarcinoma.
* The lower edge of the primary tumor is located below the peritoneal reflection or located ≤ 10 cm above the anal verge.
* Clinical stage: T3-4NanyM0 or T1-2N+M0.
* Adequate bone marrow function as evidenced by: Absolute neutrophil count (ANC) ≥1.5×10^9/L, Platelet count ≥100×10^9/L, Hemoglobin (Hb) ≥90 g/L.
* Adequate hepatic function as evidenced by: Total bilirubin ≤1.5 × upper limit of normal (ULN), Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN, Serum albumin ≥3 g/dL.
* Adequate renal function as evidenced by: Serum creatinine (Cr) ≤1.5 × ULN or creatinine clearance ≥60 mL/min.
* Be willing to undergo UGT1A1 gene testing and UGT1A1 genotype of *1*1 or *1*28.
* Accept the neoadjuvant chemoradiotherapy protocol of this study and sign the informed consent.

Exclusion Criteria:

* Any other malignancy within 5 years, with the exception of cured in-situ carcinoma or basal cell carcinoma etc.
* Active, uncontrolled bacterial, viral, or fungal infections that require systemic treatment.
* Active HIV infection.
* Combined with uncontrollable systemic diseases.
* History of allergy or hypersensitivity to drug or any of their excipients.
* Any clinical indicators indicating contraindications to radiotherapy/chemotherapy and surgery.
* Use of strong inhibitors or inducers of CYP3A, CYP2C8 and UGT1A1.
* Pregnant or breastfeeding women, or subjects of childbearing age who refuse contraception.
* Patients with poor cognitive abilities who are unable to answer questions, fill out questionnaires, or have mental disorders.
* Patients who do not meet the inclusion criteria; patients who meet the inclusion criteria but are not suitable to participate in this trial judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response | 1 week after sugery
  Defined as the proportion of patients who have achieved pathologic complete response.

SECONDARY OUTCOMES:
clinical complete response | up to 30 weeks
  Defined as the proportion of patients who have achieved clinical complete response.
Major Pathologic Response | 1 week after sugery
  Defined as the proportion of patients who have achieved major pathologic response
Objective Response Rate | through study completion，an average of 3 year
  Defined as the proportion of patients who achieved complete response (CR) and partial response (PR) according to RECIST v1.1.
Anal Sphincter Retention Rate | 1 week after sugery
  Defined as the proportion of patients who retain anal sphincter
R0 resection rate | 1 week after sugery
  Defined as the proportion of patients who have achieved R0 resection.
3-year Local Recurrence Free Survival Rate | 3 years
  Defined as the proportion of patients who are not local recurrence or death at 3 years after enrollment.
3-year Progress Free Survival Rate | 3 years
  Defined as the proportion of patients who are not progress or death at 3 years after enrollment.
3-year Overall Survival Rate | 3 years
  Defined as the proportion of patients who are alive at 3 years after enrollment.
Incidence of adverse events | 7 months
  Use NCI-CTCAE version 5.0 for classification and grading.

CONTACTS AND LOCATIONS:
Overall Officials: Fengpeng Wu, Professor, Principal Investigator — Hebei Medical University Fourth Hospital
Locations (1):
- Hebei Medical University Fourth Hospital, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No